CLINICAL TRIAL: NCT04424160
Title: Effects of Intrauterine Platelet Rich Plasma (PRP) on Endometrium and Pregnancy Rates in Patients With Suboptimal Endometrium Undergoing Frozen Embryo Transfer
Brief Title: Effects of Platelet Rich Plasma on Endometrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Baskent University (Other)
Responsible Party: Principal Investigator, Bulent Tiras, Prof., Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA20/23
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Asherman Syndrome
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Intervention Model Description: Intrauterine platelet rich plasma will be injected in the endometrial region via the vaginal route after the cessation of menstrual period. Approximately 20 ml of blood sample will be collected under sterile conditions, and PRP will be prepared. The same day, within 2 hours of sample preparation, PRP injection will be performed transvaginally under ultrasound guidance and under sedation anesthesia into the endometrial region of the endometrium in several positions.On the same day after the procedure, the patient will be observed in the outpatient room and will be discharged on the same day. On the second menstrual cycle after the procedure, the patients will be checked under ultrasound and will be started hormone replacement therapy for embryo transfer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endometrial PRP (Experimental): Patients in whom endometrial PRP was performed
  Interventions: Biological: PRP injection in the endometrium

INTERVENTIONS:
Biological: PRP injection in the endometrium — Within 5 days after the cessation of menstrual period, endometrial PRP procedure will be planned. Approximately 20 ml of blood sample will be collected under sterile conditions, and PRP will be prepared. The same day, within 2 hours of sample preparation, PRP injection will be performed transvaginally under ultrasound guidance and under sedation anesthesia into the endometrial region of the endometrium in several positions.On the same day after the procedure, the patient will be observed in the outpatient room and will be discharged on the same day.

SUMMARY:
Intrauterine platelet rich plasma will be injected in the endometrial region via the vaginal route after the cessation of menstrual period. The endometrial thickness will be assessed under ultrasound and hormone replacement will be started. As the endometrial thickness reaches adequate thickness during ultrasound follow-up, embryo transfer will be performed.

DETAILED DESCRIPTION:
Intrauterine platelet rich plasma will be injected in the endometrial region via the vaginal route after the cessation of menstrual period. In the second menstrual period following the PRP injection, the endometrial thickness will be assessed under ultrasound and hormone replacement will be started. As the endometrial thickness reaches adequate thickness during ultrasound follow-up, embryo transfer will be performed. Pregnancy test results will be recorded and followed.

ELIGIBILITY:
Inclusion Criteria:

* Women in whom cycle was cancelled due to an endometrial thickness <7 mm when progesterone start was planned in patients undergoing frozen embryo transfer with hormone replacement therapy
* Women with a history of Asherman syndrome, but no obvious intrauterine adhesion in the last hysteroscopic procedure;
* Women who have at least 2 frozen good-quality embryos.

Exclusion Criteria:

* Women with any other known cause of implantation failure, such as poor embryo quality, or congenital uterine anomalies, endometrial polyp or fibroid,
* Previous diagnosis of any malignancy,
* Anticoagulant use for which plasma infusion is contraindicated,

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All infertile women desiring pregnancy
Enrollment: 150 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness during hormone replacement therapy | 2-10 months
  To measure endometrial thickness assessed by ultrasound during hormone replacement therapy for endometrial preparation in frozen-thawed cycles

SECONDARY OUTCOMES:
Pregnancy outcomes after frozen-thawed embryo transfer | 2-10 months
  To assess pregnancy rates by beta-human chorionic gonadotropin and ultrasound after frozen-thawed embryo transfer cycles

CONTACTS AND LOCATIONS:
Overall Officials: Hulusi Bulent Zeyneloglu, Prof, Principal Investigator — Baskent University Departments of Obstetrics and Gynecology; Yigit Cakiroglu, Assoc.Prof., Study Director — Acibadem University
Locations (1):
- Acıbadem Maslak Hospital IVF Unit, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang Y, Li J, Chen Y, Wei L, Yang X, Shi Y, Liang X. Autologous platelet-rich plasma promotes endometrial growth and improves pregnancy outcome during in vitro fertilization. Int J Clin Exp Med. 2015 Jan 15;8(1):1286-90. eCollection 2015. PMID 25785127
- [Result] Tandulwadkar SR, Naralkar MV, Surana AD, Selvakarthick M, Kharat AH. Autologous Intrauterine Platelet-Rich Plasma Instillation for Suboptimal Endometrium in Frozen Embryo Transfer Cycles: A Pilot Study. J Hum Reprod Sci. 2017 Jul-Sep;10(3):208-212. doi: 10.4103/jhrs.JHRS_28_17. PMID 29142450
- [Result] Zadehmodarres S, Salehpour S, Saharkhiz N, Nazari L. Treatment of thin endometrium with autologous platelet-rich plasma: a pilot study. JBRA Assist Reprod. 2017 Feb 1;21(1):54-56. doi: 10.5935/1518-0557.20170013. PMID 28333034
- [Result] Chang Y, Li J, Wei LN, Pang J, Chen J, Liang X. Autologous platelet-rich plasma infusion improves clinical pregnancy rate in frozen embryo transfer cycles for women with thin endometrium. Medicine (Baltimore). 2019 Jan;98(3):e14062. doi: 10.1097/MD.0000000000014062. PMID 30653117
- [Derived] Cakiroglu Y, Tohma YA, Yuceturk A, Karaosmanoglu O, Aslan IO, Kopuk SY, Korun ZEU, Yazicioglu C, Zeyneloglu HB, Tiras B. A novel technique- subendometrial autologous platelet rich plasma injection in patients with unresponsive thin endometrium undergoing frozen-thawed embryo transfer: a prospective cohort study. BMC Pregnancy Childbirth. 2025 Mar 17;25(1):297. doi: 10.1186/s12884-025-07400-x. PMID 40098101